CLINICAL TRIAL: NCT06668272
Title: Small Changes Clinical Weight Loss Trial
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Leah Whigham, Associate Professor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HSC-SPH-24-0430
Record Dates: First submitted 2024-10-30; First posted 2024-10-31 (Actual); Last update posted 2024-10-31 (Actual); Status verified 2024-10

CONDITIONS: Obesity
Keywords: Small Changes; weight loss
MeSH Terms: conditions — Obesity; Weight Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Small Changes program (Experimental)
  Interventions: Behavioral: Small Changes program
- Standard behavioral therapy for weight loss (Active Comparator)
  Interventions: Behavioral: Standard behavioral therapy for weight loss

INTERVENTIONS:
Behavioral: Small Changes program — Participants will be asked to track their compliance with their Small Changes diet plan using a simple checklist record . Participants will be asked to follow their diet plan every day. They are encouraged to create a diet plan that is as close to their current diet as possible. Meal options include make-from-scratch recipes, quick "grab-and-go" options,and restaurant options. There may be some time involved in learning the recipes and the routine of their new diet. It also may alter their grocery spending and habits somewhat
  Arms: Small Changes program
Behavioral: Standard behavioral therapy for weight loss — Participants will be provided guidance on cutting and counting calories, setting goals, reading labels, and portion sizes.
  Arms: Standard behavioral therapy for weight loss

SUMMARY:
The purpose of this study is to assess the effectiveness of the Small Changes program in facilitating weight loss and to assess treatment effects on body composition, blood markers of metabolic health, and blood pressure, and to assess attrition and compliance

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index greater than or equal to 25
* Stable weight with less than a 5% body weight change in the past 3 months.
* Willingness and ability to follow a written dietary plan.
* Ambulatory and capable of attending bi-weekly in-person and phone appointments.
* Must reside in the geographic area for the duration of the 12-week study.
* Clearance for weight loss by their health care provider.

Exclusion Criteria:

* Pregnant or lactating.
* Acute medical conditions such as kidney disease, liver disease, pancreatitis, or cancer.
* A history of bariatric surgery or gastrointestinal resection.
* Current use of anti-obesity medications or diabetes medications, such as Glucagon-like peptide-1 receptor agonists (GLP-1RAs), that induce weight loss.
* A history of commercial weight loss program participation within the last six months.
* A history of anorexia nervosa or other eating disorders.
* A history of anxiety or depression.
* Extreme dietary restrictions or allergies that limit the ability to follow the weight loss plan.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2024-11-01 (Estimated); Primary Completion 2025-11-01 (Estimated); Study Completion 2025-11-01 (Estimated)

PRIMARY OUTCOMES:
Change in weight | Baseline,12 weeks

SECONDARY OUTCOMES:
Change in Hemoglobin A1C levels | Baseline, 12 weeks
Change in triglycerides levels | Baseline, 12 weeks
Change in total cholesterol levels | Baseline, 12 weeks
Change in HDL cholesterol levels | Baseline, 12 weeks
Change in fasting blood glucose levels | Baseline, 12 weeks
Change in lean body mass | baseline, week 4, week 8, week 12
Change in fat mass | baseline, week 4, week 8, week 12
Compliance as measured by the percentage of meals that follow the diet plan as reported in a daily food log | From baseline to week 12
Attrition as assessed by number of participants that complete the study | week 12

CONTACTS AND LOCATIONS:
Overall Officials: Leah Whigham, PhD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (2):
- United States (2):
  - The University of Texas Health Science Center at Houston, Houston, Texas
  - Texas Tech University, Lubbock, Texas

IPD SHARING:
Plan to Share IPD: No